CLINICAL TRIAL: NCT05933265
Title: A Phase 1/2 Dose Escalation and Cohort Expansion Study of LP-184 in Patients With Advanced or Metastatic Solid Tumors
Brief Title: Study of LP-184 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lantern Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LTRN184-1AST23-1
Record Dates: First submitted 2023-06-23; First posted 2023-07-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Advanced Solid Tumor; Metastatic Solid Tumor; GBM; TNBC - Triple-Negative Breast Cancer; NSCLC; Pancreatic Adenocarcinoma; DDR Gene Mutation
Keywords: LP-184; Phase 1; Lantern Pharma; Cancer; DNA damage repair
MeSH Terms: conditions — Neoplasm Metastasis; Triple Negative Breast Neoplasms; Neoplasms | interventions — Spironolactone; olaparib

STUDY DESIGN:
Intervention Model Description: BOIN Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Master Protocol (Experimental): A phase 1/2 dose escalation and cohort expansion study of LP-184 in patients with advanced or metastatic solid tumors. A BOIN design will be used to evaluate the safety of LP-184, determine the MTD, and identify the RP2D. Patients who meet all eligibility criteria will be enrolled to receive treatment with LP-184 at a dose determined based on the available cohort at the time of each patient's enrollment. Patients will receive LP-184 infusion during Day 1 and Day 8 of each 21-day cycle, for a minimum of two cycles.
  Interventions: Drug: LP-184
- Supplement A (Experimental): Phase 1b/2 Expansion cohort of participants with triple negative breast cancer (TNBC), non-small cell lung cancer (NSCLC), pancreatic adenocarcinoma (PDAC) or other solid tumours with known DDR genomic alterations to determine the optimal dose/RP2D and to obtain preliminary estimates of clinical activity.
  Interventions: Drug: LP-184
- Supplement B (Experimental): Phase 1b/2 Expansion cohort of participants with recurrent GBM to evaluate the safety, pharmacokinetics and preliminary anti-tumour activity of LP-184 alone and in combination with spironolactone.
  Interventions: Drug: LP-184; Drug: Spironolactone
- Supplement C (Experimental): Phase 1b/2 Expansion cohort of participants with Hormone Receptor (HR)-Negative and HER2-Negative Breast Cancer (TNBC) to evaluate the safety, tolerability and clinical activity of LP-184 in combination with olaparib
  Interventions: Drug: LP-184; Drug: Olaparib

INTERVENTIONS:
Drug: LP-184 — LP-184 is a small molecule alkylating agent causing tumor cell death through DNA damage.
Drug: Spironolactone — A competitive mineralocorticoid receptor antagonist that inhibits aldosterone-dependent sodium reabsorption/ potassium excretion and lowering blood pressure, as well as degrades the transcription coupled nucleotide excision repair protein ERCC3 to impair DNA repair.
  Arms: Supplement B
Drug: Olaparib — A poly (ADP-ribose) polymerase (PARP) inhibitor that impairs homologous recombination (HR) dependent DNA damage repair by trapping PARP1/2 on DNA, leading to synthetic lethality in BRCA1/2-deficient cells.
  Arms: Supplement C

SUMMARY:
The primary objective of this study is to evaluate the safety, tolerability, MTD and RP2D of LP-184 in patients with advanced solid tumors who have relapsed from or are refractory to standard therapy or for whom no standard therapy is available. The secondary objectives are to characterize the PK of LP-184 and its metabolites in plasma and assess clinical activity of LP-184.

Participants will receive LP-184 infusion during Day 1 and Day 8 of each 21-day cycle, for a minimum of two cycles. Patients will be monitored for safety, PK, and clinical activity

DETAILED DESCRIPTION:
Patients who meet all eligibility criteria will be enrolled to receive treatment with LP-184 at a dose determined based on the available cohort at the time of each patient's enrollment. Patients will receive LP-184 infusion during Day 1 and Day 8 of each 21-day cycle, for a minimum of two cycles. Patients will be monitored for safety, PK, and clinical activity. Dose escalation is planned with minimum of 3 patient cohorts (starting at dose level 1). After selection of the maximum tolerated dose (MTD), additional patients will be enrolled at two dose levels, including the MTD, as determined by the Safety Review Committee, until at least 10 patients each are treated at each dose to determine the recommended phase 2 dose.

ELIGIBILITY:
Patient Inclusion Criteria:

1. ≥18 years of age at the time of consent
2. Provided signed written ICF and voluntary consent prior to any mandatory study-specific procedures, sampling, and analyses.
3. Have a histologically or cytologically documented advanced solid tumor that has relapsed from or is refractory to standard treatment, or for which no standard treatment is available.

   Note: patients with certain tumor types such as those with relatively high prevalence of DDR gene alterations and/or PTGR1 over expression (e.g., triple negative breast cancer, lung, prostate, ovarian, pancreatic, bladder, and GBM) may be preferentially enrolled in Phase 1a.
4. ECOG performance status 0-1 or Karnofsky performance scale >60 for GBM patients.
5. Patients must have measurable disease per RECIST 1.1 or RANO 2.0 criteria as applicable.

   Note: patients without measurable disease may be eligible, following discussion with the investigator and the sponsor, if the patient presents with non-measurable but evaluable disease of any size unequivocally attributable to advanced solid tumor.
6. Patients must have life expectancy >3 months.
7. Adequate organ function at screening defined as:

   Liver Function
   * AST, ALT ≤3 x ULN or <5 x ULN in cases of documented liver metastases or involvement of liver in the disease process.
   * Total serum bilirubin ≤1.5 x ULN or <5 x ULN if secondary to Gilbert's syndrome or documented liver metastases or involvement of liver in the disease process.

   Renal Function
   * Serum creatinine clearance ≥60 mL/min either measured or calculated using standard Cockcroft-Gault formula.
   * Serum electrolyte (potassium, calcium, and magnesium) levels within the normal reference range (may be supplemented according to institutional standard).

   Bone Marrow Function:
   * ANC ≥1500/μL.
   * Hemoglobin ≥8 g/dL (The use of transfusion or other intervention to achieve hemoglobin ≥8 g/dL is acceptable. For those patients undergoing RBC transfusion, hemoglobin must be evaluated at least 14 days after the last RBC transfusion).
   * Platelet count ≥100,000/μL (assessed ≥7 days following last platelet transfusion in patients with thrombocytopenia requiring platelets).

   Blood clotting function:

   - INR and aPTT ≤1.5 x ULN. Study patients on therapeutic doses of anticoagulation medication must have INR and/or aPTT ≤ the upper limit of the therapeutic range for intended use.
8. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 3 days of first dose of LP-184. A woman is of child-bearing potential unless she:

   * has had a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy;
   * is age ≥60 years and is amenorrhoeic; or
   * is age <60 years and has been amenorrhoeic for ≥12 months (including no irregular menses or spotting) in the absence of any medication which induces a menopausal state and has documented ovarian failure by serum estradiol and follicle-stimulating hormone levels within the institutional laboratory postmenopausal range).
9. WOCBP or must agree to use highly effective contraceptive methods and avoid egg donation during the study treatment and for 6 months after the last dose of LP-184.
10. Men of reproductive potential agree to use highly effective contraceptive methods and avoid sperm donation during the study treatment and for 3 months after the last dose of LP-184. A man is of child-producing potential unless he has had a bilateral vasectomy with documented aspermia or a bilateral orchiectomy.
11. Is willing to provide archived samples (blocks and/or slides) for comprehensive DDR genomic analyses and/or PTGR1 expression profiling and/or other genomic alterations if the patient has a PR/CR.
12. Regarding brain metastases, based on screening contrast brain MRI, patients must have 1of the following:

    * No evidence of brain metastases
    * Untreated brain metastases not requiring immediate local therapy. For patients with untreated CNS lesions >2.0 cm on screening contrast brain MRI, discussion with and approval from the Medical Monitor is required prior to enrollment.
    * Previously treated brain metastases that are either stable for at least 4 weeks since last treatment or progressed since prior local CNS therapy and not requiring immediate re-treatment with local therapy in the opinion of the investigator.

Patient Exclusion Criteria:

1. Exposure to anti-cancer therapy within 2 weeks or within at least 5 half-lives of the anticancer agent whichever is shorter; or 4 weeks from any biologics/immunotherapies or any investigational therapy prior to the first dose of LP-184.

   Note: Low dose steroids (oral prednisone or equivalent ≤20 mg/day, except patients with GBM), localized non-CNS radiotherapy, previous hormonal therapy with luteinizing hormone-releasing hormone agonists for prostate cancer and treatment with bisphosphonates and RANKL inhibitors are not criteria for exclusion if such therapy has not been changed within 4 weeks before LP-184 treatment.
2. Any history of retinopathy and/or macular degeneration (without specifications or grades).
3. Has received radiation within 4 weeks of Cycle 1 Day 1. Unless the tumor at the site of treatment continues to increase in size after the patient has completed radiotherapy treatment.
4. Infection requiring antibiotics, antivirals, or antifungals within 1 week prior to first dose of study drug, unless such infection is adequately controlled (defined as exhibiting no ongoing signs/symptoms related to the infection and with clinical improvement). In the case of prophylactic use of these agents, discussion with the Medical Monitor is required prior to enrollment.
5. Hepatitis B and/or hepatitis C infection (as detected by positive testing for hepatitis B surface antigen [HbsAg] or antibody to hepatitis C virus with confirmatory testing) or known seropositivity for or history of active viral infection with human immunodeficiency virus (HIV).
6. Are pregnant or breastfeeding. (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
7. Have clinically significant cardiac disease including:

   * New York Heart Association Class IV heart failure.
   * Myocardial infarction or stroke ≤3 months prior to the first dose of LP-184.
   * Unstable angina within ≤12 weeks prior to the first dose of LP-184 unless the underlying disease has been corrected by procedural intervention e.g., stent, bypass.
   * Severe aortic stenosis.
   * Uncontrolled arrhythmia. Sponsor approval of patients with arrhythmia is required.
   * QTc >470 ms by Fredericia criteria.
   * Congenital long QT syndrome, or a QT interval corrected by Fridericia's formula (QTcF) >470 ms (average of triplicate ECGs) at Screening and/or on Cycle 1 Day 1 (pre-dose) except for a documented bundle branch block or unless secondary to pacemaker. In the case of a documented bundle branch block or a pacemaker, discussion with the medical monitor is required prior to enrollment.
8. Have clinically significant AEs that have not returned to baseline or ≤Grade 1 based on NCI-CTCAE prior to first dose of study drug, unless approved by the sponsor. Patients with chronic Grade 2 toxicities may be eligible per the discretion of the investigator and sponsor (e.g., Grade 2 chemotherapy-induced neuropathy, alopecia, or hypothyroidism from prior immunotherapy treatment).
9. Have had major surgery (requiring general anesthesia) within ≤4 weeks of first dose of LP-184.
10. Have any other serious medical condition which, in the opinion of the investigator, would preclude the patient from study participation.
11. Have clinically active brain metastases, defined as untreated and symptomatic, or requiring therapy with steroids at a dose > 2 mg of dexamethasone or equivalent or anticonvulsants to control associated symptoms. Patients with treated brain metastases that are no longer symptomatic and who require no treatment with steroids may be included in the study if they have recovered from the acute toxic effect of radiotherapy. A minimum of 4 weeks must have elapsed between the end of whole brain radiotherapy and study enrollment (1 week for stereotactic radiotherapy).
12. For patients with suspected or known CNS metastatic disease, based on screening brain MRI, patients must not have:

    Any untreated brain lesions >2.0 cm in size unless Medical Monitor approved enrollment.

    Ongoing use of systemic corticosteroids for control of symptoms of brain metastases at a total daily dose of >2 mg of dexamethasone (or equivalent).

    Patients on a chronic stable dose of ≤2 mg total daily of dexamethasone (or equivalent) are eligible with discussion and approval by the medical monitor. (Note: this is not applicable to patients with GBM).

    Any brain lesion thought to require immediate local therapy, including (but not limited to) a lesion in an anatomic site where an increase in size or possible treatment-related edema may pose a risk to the patient (e.g., brain stem lesions). Patients who underwent local treatment for such lesions identified by screening contrast brain MRI may still be eligible based on criteria described under CNS inclusion criteria described above.

    • Known or suspected leptomeningeal disease as documented by the investigator.
13. Male patients with partners currently pregnant, or male patients able to father children, and female patients of childbearing potential who are unwilling or unable to use highly effective methods of contraception as outlined in this protocol for the duration of the study and for at least 3 months (male) or 6 months (female) after last dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2023-06-09 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-09-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of LP-184 assessed by the incidence and severity of all adverse events graded by CTCAE v5.0 | 12 months
To determine the MTD of LP-184 based on all available safety (graded by CTCAE v5.0) and PK data. | 12 months
To determine the RP2D of LP-184 based on all available safety (graded by CTCAE v5.0), PK, PD and efficacy data | 12 months

SECONDARY OUTCOMES:
To characterize the PK of LP-184 and its metabolites in plasma by assessing the area under the plasma concentration versus time curve (AUC). | Blood samples for PK analysis collected at multiple time points during cycle 1 (each cycle is 21 days)
To characterize the PK of LP-184 and its metabolites in plasma by assessing the peak plasma concentration (Cmax) | Blood samples for PK analysis collected at multiple time points during cycle 1 (each cycle is 21 days)
To characterize the PK of LP-184 and its metabolites in plasma by assessing the time to peak plasma concentration (Tmax) | Blood samples for PK analysis collected at multiple time points during cycle 1 (each cycle is 21 days)
To characterize the PK of LP-184 and its metabolites in plasma by assessing the amount of time required for the drug concentration in plasma to be reduced to exactly half its starting concentration (half-life, t1/2) | Blood samples for PK analysis collected at multiple time points during cycle 1 (each cycle is 21 days)
To characterize the PK of LP-184 and its metabolites in plasma by assessing the apparent volume of distribution at steady state after non-intravenous administration (Vss/F) | Blood samples for PK analysis collected at multiple time points during cycle 1 (each cycle is 21 days)
To assess the clinical activity of LP-184. Overall response rates defined as percentage of patients with CR or PR per RECIST 1.1 or RANO 2.0 criteria in Gliomas | Tumor imaging is obtained every 6 weeks or 2 cycles (each cycle being 21 days long) for the first 5 cycles and every 12 weeks or 4 cycles unless increased frequency is clinically indicated up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Reggie Ewesuedo, MD, Study Director — Lantern Pharma Inc.
Locations (9):
- United States (9):
  - Highlands Oncology Group, Springdale, Arkansas
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - Northwest Oncology & Hematology, Rolling Meadows, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Norton Healthcare, Inc., Louisville, Kentucky
  - John Hopkins - The Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UT Health Science Center San Antonio, San Antonio, Texas
  - START Mountain Region, West Valley City, Utah

IPD SHARING:
Plan to Share IPD: No